CLINICAL TRIAL: NCT02906371
Title: A Two Cohort Pilot Study of the Tocilizumab Optimization Timing for CART19 Associated Cytokine Release Syndrome (CRS) Management in Pediatric Patients With CD19 Expressing Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia (ALL)
Brief Title: Study of the Tocilizumab Optimization Timing for CART19 Associated Cytokine Release Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16CT022, 825445
Record Dates: First submitted 2016-08-29; First posted 2016-09-20 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Lymphoblastic Leukemia, Acute, Childhood
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tocilizumab high tumor burden (Active Comparator): This is a two cohort, open-label, pilot study to describe the efficacy of administration timing of tocilizumab on CART19 (CTL019) associated CRS safety events in pediatric patients with CD19 expressing relapsed and refractory B-cell acute lymphoblastic leukemia with high pre-infusion tumor burden following redirected autologous T cells transduced with the anti-CD19 lentiviral vector (CART19/CTL019).
  Interventions: Drug: Tocilizumab; Biological: CART 19
- Tocilizumab low tumor burden (Active Comparator): This is a two cohort, open-label, pilot study to describe the efficacy of administration timing of tocilizumab on CART19 (CTL019) associated CRS safety events in pediatric patients with CD19 expressing relapsed and refractory B-cell acute lymphoblastic leukemia with low pre-infusion tumor burden following redirected autologous T cells transduced with the anti-CD19 lentiviral vector (CART19/CTL019).
  Interventions: Drug: Tocilizumab; Biological: CART 19

INTERVENTIONS:
Drug: Tocilizumab — Patients with ≥ 40% blasts in the bone marrow at pre-infusion will be enrolled in the early tocilizumab cohort and will follow early CRS treatment algorithm.
  Other Names: high tumor burden
  Arms: Tocilizumab high tumor burden
Drug: Tocilizumab — Patients with ˂ 40% blasts in the bone marrow at pre-infusion (~ Day -5 to -1) will follow the standard CRS Rx algorithm
  Other Names: low tumor burden
  Arms: Tocilizumab low tumor burden
Biological: CART 19 — CART-19 cells transduced with a lentiviral vector to express either anti-CD19ζ scFv TCRζ:41BB, administered by i.v. injection using an intra-patient dose escalation approach: 10% on day 0, 30% on day 1 with a total dose goal of ~1.5 x107 - 5 x109 (~3x105 - 1x108/kg) T cells.

SUMMARY:
This is a two cohort, open-label, pilot study to describe the efficacy of administration timing of tocilizumab on CART19 (CTL019) associated cytokine release syndrome safety events in pediatric patients with CD19 expressing relapsed and refractory B-cell acute lymphoblastic leukemia with high versus low pre-infusion tumor burden following redirected autologous T cells transduced with the anti-CD19 lentiviral vector (CART19/CTL019).

DETAILED DESCRIPTION:
The duration of active protocol intervention is approximately 12-15 months from the screening visit. The protocol will require approximately 12-18 months to complete enrollment.Approximately 39 enrolled patients to reach at least 35 infused patients, with the ultimate goal of 15 patients in the high tumor burden cohort (Cohort A). Inclusion criteria are designed to include pediatric patients aged 1-24 years with CD19 expressing relapsed/refractory B-cell acute lymphoblastic leukemia (ALL).Tocilizumab will be given once to high disease burden patients, and then the patients will be managed for CRS as per the standard algorithm (including subsequent tocilizumab, if needed).

Two cohorts are defined based upon pre-infusion high versus low tumor burden; with the high tumor burden cohort (high risk of severe CRS) to receive earlier administration of tocilizumab for CRS management and the low tumor burden cohort (low risk of severe CRS) to receive standard timing of tocilizumab for CRS

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form must be obtained prior to any study procedure. Labs, marrows or other procedures obtained during routine clinical care may be used for eligibility if obtained within the protocol required windows.
2. Relapsed or refractory B-cell ALL:

   1. 2nd or greater marrow relapse OR
   2. CNS relapse OR
   3. Any relapse after allogeneic hematopoietic stem cell (SCT) transplant and ≥ 4 months from SCT at enrollment OR
   4. Any relapse after CAR-modified T cell therapy OR
   5. Refractory disease defined as having not achieved an MRD-negative CR after ≥ 2 chemotherapy regimens/cycles (1 cycle for relapsed patients) OR
   6. Patients with Ph+ ALL are eligible if they are intolerant to or have failed tyrosine kinase inhibitor therapy OR
   7. Ineligible for allogeneic SCT because of:

      * Comorbid disease
      * Other contraindications to allogeneic SCT conditioning regimen
      * Lack of suitable donor
      * Prior SCT
      * Declines allogeneic SCT as the therapeutic option after documented discussion, with expected outcomes, about the role of SCT with a bone marrow transplant (BMT) physician not part of the study team
   8. Patients with B lymphoblastic lymphoma will be eligible if they meet one of the above criteria OR:

      * 2nd or greater relapse OR
      * Refractory disease defined as having not achieved CR with frontline therapy or after 1 cycle of reinduction therapy for relapsed patients
   9. Patients with prior or current history of CNS3 disease will be eligible if CNS disease is responsive to therapy (at infusion, must meet criteria in Section 5.3)
3. Documentation of CD19 tumor expression in bone marrow, peripheral blood, CSF, or tumor tissue by flow cytometry at relapse (or a recent sample in the case of refractory disease). If the patient has received CD19-directed therapy (i.e. blinatumomab), then the flow cytometry should be obtained after this therapy to show CD19 expression.
4. Adequate organ function defined as:

   1. A serum creatinine based on age/gender as follows:

      Maximum Serum Creatinine (mg/dL)

      Age Male Female
      * 1 to < 2 years 0.6 0.6
      * 2 to < 6 years 0.8 0.8
      * 6 to < 10 years 1.0 1.0
      * 10 to < 13 years 1.2 1.2
      * 13 to < 16 years 1.5 1.4
      * ≥ 16 years 1.7 1.4
   2. ALT ≤500 U/L
   3. Bilirubin ≤2.0 mg/dl
   4. Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea, pulse oximetry > 92% on room air; DLCO ≥ 40% (corrected for anemia) if PFTs are clinically appropriate as determined by the treating investigator
   5. Left Ventricular Shortening Fraction (LVSF) ≥ 28% or Ejection Fraction (LVEF) ≥ 40% confirmed by ECHO, or adequate ventricular function documented by a scan or a cardiologist.
5. Evidence of disease by standard morphologic or MRD criteria. A clinical marrow or tissue biopsy showing disease may be performed at enrollment or within 12 weeks of enrollment. Presence of marrow disease not required for CNS disease or lymphoblastic lymphoma patients.
6. Age 1-29 years. Patients ages 24-29 years are eligible if their original leukemia diagnosis was prior to age 21.
7. Adequate performance status (Lansky or Karnofsky score ≥50).
8. Subjects of reproductive potential must agree to use acceptable birth control methods, as described in protocol Section 4.3.

Exclusion Criteria:

1. Active hepatitis B or active hepatitis C.
2. HIV Infection.
3. Active acute or chronic graft-versus-host disease (GVHD) requiring systemic therapy.

5. CNS3 disease that is progressive on therapy, or with CNS parenchymal lesions that might increase the risk of CNS toxicity.

6. Pregnant or nursing (lactating) women. 8. Uncontrolled active infection.

Ages: 1 Year to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2016-08; Primary Completion 2020-03-11 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
the frequency of grade 4 CRS | from day 1 to 1 year
  Frequency of CRS grade 4

SECONDARY OUTCOMES:
tumor response | day 28
  Frequency of CR with minimal residual disease negative bone marrow at day 28 and duration of remission

OTHER OUTCOMES:
CART19 cellular kinetics | from day -1 to year 1
  Peak plasma concentration (Cmax) of CART19 cellular kinetic
Number of days in ICU | from day 0 through year one.
Frequency of major medical interventions | from day 0 through year one.
CART19 cellular kinetics | from day -1 through year 1
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan A Grupp, MD,PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kadauke S, Myers RM, Li Y, Aplenc R, Baniewicz D, Barrett DM, Barz Leahy A, Callahan C, Dolan JG, Fitzgerald JC, Gladney W, Lacey SF, Liu H, Maude SL, McGuire R, Motley LS, Teachey DT, Wertheim GB, Wray L, DiNofia AM, Grupp SA. Risk-Adapted Preemptive Tocilizumab to Prevent Severe Cytokine Release Syndrome After CTL019 for Pediatric B-Cell Acute Lymphoblastic Leukemia: A Prospective Clinical Trial. J Clin Oncol. 2021 Mar 10;39(8):920-930. doi: 10.1200/JCO.20.02477. Epub 2021 Jan 8. PMID 33417474
- See also: Related Info — http://www.chop.edu/service/oncology/pediatric-cancer-research/cart-19-trial.html